CLINICAL TRIAL: NCT03040206
Title: Multicenter Study to Assess the Prognostic Significances of NCCN-IPI and Post-treatment PET Results in Patients With Newly Diagnosed Nodal PTCL
Brief Title: Risk Stratification of Nodal PTCL
Status: Completed | Type: Observational
Sponsor: Chonbuk National University Hospital (Other)
Collaborators: Chonnam National University Hospital (Other); Kyungpook National University Hospital (Other); Keimyung University Dongsan Medical Center (Other); Korea University Anam Hospital (Other); Korea University Guro Hospital (Other); Dong-A University Hospital (Other); Pusan National University Hospital (Other); Yeungnam University Hospital (Other); Inje University (Other); Chungnam National University Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ho-Young Yhim, Assistant professor, Chonbuk National University Hospital
Other Study IDs: nodal PTCL
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Peripheral T-Cell Lymphoma, Not Otherwise Specified; Angioimmunoblastic T-cell Lymphoma; Anaplastic Large Cell Lymphoma, ALK-negative
MeSH Terms: conditions — Lymphoma, T-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nodal PTCL: 1. newly-diagnosed, pathologically-proven nodal PTCLs (PTCL, NOS; Angioimmunblastic T-cell lymphoma; anaplastic large cell lymphoma [ALCL], anaplastic lymphoma kinase [ALK]-negative) between January 1, 2005 and Jun 30, 2016
  2. initially treated with curative intent
  3. Standard PET or PET-CT data available at the time of diagnosis and at the end of primary treatment

SUMMARY:
This study is to investigate the prognostic significance of enhanced International Prognostic Index (NCCN-IPI) and post-treatment PET results in patients with newly diagnosed nodal peripheral T-cell lymphoma (PTCL), and establish a risk stratification model for nodal PTCL patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with nodal PTCLs (PTCL, NOS; Angioimmunblastic T-cell lymphoma; anaplastic large cell lymphoma [ALCL], anaplastic lymphoma kinase [ALK]-negative)
* Patients diagnosed with between January 1, 2004 and April 30, 2016
* initially treated with curative intent
* Patients with standard 18F-fluorodeoxyglucose (FDG) PET or PET-CT data at the time of diagnosis and at the end of primary treatment

Exclusion Criteria:

* Patients diagnosed with extranodal PTCLs, including followings (extranodal NK/T-cell lymphoma, nasal type; enteropathy-associated T-cell lymphoma; hepatosplenic T-cell lymphoma; subcutaneous panniculitis-like T-cell lymphoma; EBV-positive T-cell lymphoproliferative childhood disorders, and primary cutaneous lymphomas)
* Patients with ALCL-ALK+
* Patients who do not have 18F-FDG PET or PET-CT data either at diagnosis or at the end of treatment available for review

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed, pathologically prove nodal PTCL (PTCN-NOS; AITL; ALCL, ALK-negative)
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 5 year
  Time between the date of diagnosis and any kinds of death or disease relapse/progrression

SECONDARY OUTCOMES:
overall survival | 5 year
  Time between the date of diagnosis and any kinds of death

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Young Yhim, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk Nationla University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No